CLINICAL TRIAL: NCT01178138
Title: Monoamine Antagonist Therapies for Methamphetamine Abuse Prazosin
Acronym: MATMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 110371; 1R01DA026916-01 (NIH)
Record Dates: First submitted 2010-08-04; First posted 2010-08-09 (Estimated); Results first posted 2014-09-08 (Estimated); Last update posted 2016-12-30 (Estimated); Status verified 2016-11

CONDITIONS: Continuous Methamphetamine Abuse
Keywords: substance abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prazosin effects on methamphetamine (Other): Randomized placebo controlled trial of prazosin effects on methamphetamine
  Interventions: Drug: Prazosin

INTERVENTIONS:
Drug: Prazosin — Prazosin or oral placebo given before methamphetamine or iv placebo to determine effects of prazosin on methamphetamine.
  Other Names: Minipress

SUMMARY:
This protocol will test the safety, effectiveness and the metabolism and action of prazosin as a potential therapy for methamphetamine abuse. This will be accomplished by performing a series of human laboratory studies. In each of these studies, the safety and effectiveness of the test medication (prazosin) in the treatment of methamphetamine effects will be determined. The study hypothesis is that prazosin will block the methamphetamine receptor function, reducing the reinforcing effects of central nervous system effects in humans.

DETAILED DESCRIPTION:
Methamphetamine (METH) use has increased in the US and worldwide in the past years. Although associated with profound medical, psychiatric, legal, and social problems, no effective medicines for METH abuse have been identified or approved for human use. It is vitally important to identify compounds that alter METH effects without increasing the risk of METH toxicity. While the brain chemical transmitter dopamine plays a major role in the pleasurable reinforcing and psychomotor stimulant effects of amphetamines, the transmitters norepinephrine and serotonin also contribute substantially to these effects. Recent evidence suggests that the functional links that exist between norepinephrine and serotonin systems may be profoundly important in METH effects and dependence. However, these neurotransmitter systems have not been tested as extensively as targets of pharmacologic interventions. Thus, the purpose of this study is to examine whether the alpha-1-b antagonist prazosin blocks the self-reported effects, cognitive performance and cardiovascular effects of METH in a dose-related manner. Subsequent protocols will test the effect of the serotonin antagonist, cyproheptadine, and the combined norepinephrine/serotonin antagonist, quetiapine. Healthy, non-treatment-seeking METH users will be recruited. They will undergo extensive prestudy medical and psychiatric screening. Twelve volunteers (ages 18-50 years; 50% female; 10% Minority) who sign the informed consent will be recruited to complete the study on prazosin.

METH-abusing volunteers will undergo 6 sessions spaced 2-3 days apart. A single oral dose of prazosin (placebo, 1 mg, or 2 mg po) will be given in a randomized, double-blind design before METH or METH placebo administration in each session. METH will be given po in a dose (20 mg) that is well-tolerated by humans but that results in easily measurable effects by itself (Cruickshank and Dyer, 2009; Sevak et al, 2009; Parrot et al, 2011). Prior to and at several time points after prazosin/placebo,METH/placebo, or prazosin/METH administrations, self-report, cognitive performance and physiologic measures will be obtained.

The studies we propose are significant as they have the potential to identify treatment medications and elucidate new mechanisms of action and desirable characteristics for future medications development. Understanding the effects of treatment drugs in the context of concomitant METH use is an essential component of identifying potential pharmacotherapies for METH dependence that 1) alters the self-reported/performance effects 2) alters the cardiovascular effects and 3) alters the concentration-effect (pharmacodynamic) relationships of METH in human METH users. Using this broad pharmacologic approach to these human laboratory studies will provide insight into the appropriate combination of positive treatment effects with minimal side effects for the ultimate development of a successful treatment for METH abuse. The results should be generalizable to METH abusers and to the development of new treatments for METH abuse that will benefit all members of society. Understanding pharmacologic interactions will lessen complications of drug abuse and provide more rapid introduction of effective new treatments into medical practice.

ELIGIBILITY:
Inclusion Criteria:

* Must be between the ages of 18-50 years (inclusive).
* Must be a current methamphetamine user, with self-reported amount of IV use being greater than the total administered in the study.
* Must have recent use confirmed by a urine toxicology screen positive for amphetamines.
* Must not be seeking treatment for methamphetamine abuse/dependence.

Exclusion Criteria:

* Ill health (major cardiovascular, renal, endocrine, hepatic disorder, to be determined by history provided by the prospective subject or laboratory evaluation as outlined below).
* Current diagnosis of other drug or alcohol physical dependence (other than nicotine or caffeine).
* History of major organic psychiatric disorder (psychosis, schizophrenia, bipolar, mania) or significant psychiatric symptoms at the time of evaluation for study participation, including suicidal ideation.
* Pregnancy, plans to become pregnant, or fertile women without adequate means of contraception.
* Present or recent use of over-the-counter or prescription psychoactive drug or drug that would have major interaction with drugs to be tested.
* Liver function tests greater than three times normal, blood urea nitrogen and creatinine outside of normal range, or thyroid function tests outside of normal range.
* EKG abnormalities including but not limited to: bradycardia (<60 bpm); prolonged corrected QT interval interval (>450 msec); Wolff-Parkinson-White syndrome; wide complex tachycardia; 2nd degree, Mobitz type II heart block; 3rd degree heart block; left or right bundle branch block.
* Medical contraindication to or prior serious adverse effects from METH or stimulants (i.e., seizures, cardiac arrest) or medical contraindication to test agents (see risks section). Significant physical or psychiatric illness which might impair the ability to safely complete the study or that might be complicated by the study drugs, including prior seizures (after age 8) or other active neurological disease or clinically significant abnormalities on physical examination or screening laboratory values.
* Current enrollment in a methamphetamine, alcohol, or other drug treatment program or current legal problems relating to METH, alcohol, or other drug use, including awaiting trial or supervision by a parole or probation officer.
* Left ventricular ejection fraction < 40% as determined in the screening echocardiogram.
* Body Mass Index >35 or <18.
* Currently trying to quit METH use.
* History of serious adverse event or hypersensitivity to methamphetamine or other study drugs
* Currently taking any medication (including highly active antiretroviral therapy for HIV) other than over-the-counter nonsteroidal anti-inflammatory medications, topical medications, inhaled asthma therapy, and over-the-counter nonsedating antihistamines.
* Any other condition the PI or staff feels will put the subject at risk for entering the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William B Gentry, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prazosin Effects on Methamphetamine: Double blind, placebo controlled study of the effect of prazosin on methamphetamine
  The order of placebo vs. active medication will be randomized.
  oral placebo and methamphetamine 20mg po: Methamphetamine 20mg po will be given 30 minutes after oral placebo.
  General Study Design. The Methamphetamine Tolerance regimen will always occur in the first study session. The medication regimen in sessions 2-6 will be randomized to one of the following five combinations of oral prazosin and iv methamphetamine.
  Session 1 (Monday) Sessions 2 - 6 (Wed, Fri, Mon, Wed, Fri).
  Oral placebo + methamphetamine (0, 15, 15 mg/70 kg) Oral placebo + methamphetamine placebo (0, 0, 0 mg/70 kg) Prazosin 1 mg po + methamphetamine placebo (0, 0, 0 mg/70 kg) Prazosin 2 mg po + methamphetamine placebo (0, 0, 0 mg/70 kg) Prazosin 1 mg po + methamphetamine (0, 15, 15 mg/70 kg) Prazosin 2 mg po + methamphetamine (0, 15, 15 mg/70 kg)
Period: Overall Study
Arm/Group | Prazosin Effects on Methamphetamine
Started | 24
Completed 6 Sessions | 1
Completed 5 Sessions | 1
Completed 3 Sessions | 1
Completed | 1
Not Completed | 23
Not completed — Lost to Follow-up | 8
Not completed — Withdrawal by Subject | 7
Not completed — Physician Decision | 8

BASELINE CHARACTERISTICS:
Population: These participants are the only ones who entered the study proper, meaning these were the only ones who received any study medications.
Groups:
- Prazosin Effects on Methamphetamine: The order of placebo vs. active medication will be randomized.
  oral placebo and methamphetamine 20mg po: Methamphetamine 20mg po will be given 30 minutes after oral placebo.
  General Study Design. The Methamphetamine Tolerance regimen will always occur in the first study session. The medication regimen in sessions 2-6 will be randomized to one of the following five combinations of oral prazosin and iv methamphetamine.
  Session 1 (Monday) Sessions 2 - 6 (Wed, Fri, Mon, Wed, Fri).
  * Oral placebo + methamphetamine (0, 15, 15 mg/70 kg)
  * Oral placebo + methamphetamine placebo (0, 0, 0 mg/70 kg)
  * Prazosin 1 mg po + methamphetamine placebo (0, 0, 0 mg/70 kg)
  * Prazosin 2 mg po + methamphetamine placebo (0, 0, 0 mg/70 kg)
  * Prazosin 1 mg po + methamphetamine (0, 15, 15 mg/70 kg)
  * Prazosin 2 mg po + methamphetamine (0, 15, 15 mg/70 kg)
Arm/Group | Prazosin Effects on Methamphetamine
Number analyzed (Participants) | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (9.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Self-report Effects of High.
Description: Visual analog scales measuring effects prazosin on methamphetamine; change in methamphetamine high. Visual analog scales allow the subject to give a rating of methamphetamine effects. For instance, how high the dose makes you . The study tested how much prazosin changed the effects of methamphetamine as measured by these visual analog scales.
  Visual analog scale is a 100 mm scale, ranging from 0 (no effect) to 100 (maximum effect).
  In each session, each subject received prazosin (1 or 2 mg) or prazosin placebo. The visual analog scale was measured. Then, one hour later, methamphetamine placebo or methamphetamine (20mg) was given and the visual analog scale was measured again.
Time Frame: 0 hr time point after prazosin and 1 hr time point after methamphetamine
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Prazosin Placebo and Methamphetamine Placebo: The order of placebo vs. active medication was be randomized to determine the how much, if any, prazosin changed the effects of methamphetamine. Visual analog scales were used to determine effects. Because only 1 subject completed the study, measures of dispersion were not reported.
Arm/Group | Prazosin Placebo and Methamphetamine Placebo | Prazosin 1 mg and Methamphetamine Placebo | Prazosin 2 mg and Methamphetamine Placebo | Prazosin 1 mg and Methamphetamine 20 mg | Prazosin 2 mg and Methamphetamine 20 mg | Prazosin Placebo and Methamphetamine 20 mg
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 1 | 3
units on a scale
  VAS baseline | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  VAS after methamphetamine | 0 (0) | 0 (0) | 0 (0) | 10 (14.1) | 15 (0) | 16.7 (15.3)

2. Primary Outcome: Heart Effects of Prazosin on Methamphetamine
Description: Heart effects of prazosin on methamphetamine;
  In each session, each subject received prazosin (1 or 2 mg) or prazosin placebo. The heart rate was measured. Then, one hour later, methamphetamine placebo or methamphetamine (20mg) was given and the heart rate was measured again.
Time Frame: 0 hr time point after prazosin and 1 hr time point after methamphetamine
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Prazosin Placebo and Methamphetamine Placebo | Prazosin 1 mg and Methamphetamine Placebo | Prazosin 2 mg and Methamphetamine Placebo | Prazosin 1 mg and Methamphetamine 20 mg | Prazosin 2 mg and Methamphetamine 20 mg | Prazosin Placebo and Methamphetamine 20 mg
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 1 | 3
beats per minute
  Heart rate baseline | 78.7 (12.5) | 74 (10.1) | 74 (0) | 75.5 (3.5) | 80 (0) | 80 (9.1)
  Heart rate methamphetamine | 72.7 (14.1) | 83.3 (10.4) | 81 (9.9) | 81.5 (9.2) | 70 (0) | 82 (6.2)

3. Primary Outcome: Blood Pressure Effects of Prazosin on Methamphetamine
Description: Blood pressure effects of prazosin on methamphetamine;
  In each session, each subject received prazosin (1 or 2 mg) or prazosin placebo. The blood pressure was measured. Then, one hour later, methamphetamine placebo or methamphetamine (20mg) was given and the blood pressure was measured again.
Time Frame: 0 hr time point after prazosin and 1 hr time point after methamphetamine
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Prazosin Placebo and Methamphetamine Placebo | Prazosin 1 mg and Methamphetamine Placebo | Prazosin 2 mg and Methamphetamine Placebo | Prazosin 1 mg and Methamphetamine 20 mg | Prazosin 2 mg and Methamphetamine 20 mg | Prazosin Placebo and Methamphetamine 20 mg
Number analyzed (Participants) | 3 | 3 | 2 | 2 | 1 | 3
mmHg
  systolic blood pressure baseline | 119.3 (14.6) | 110.3 (8.5) | 113.5 (10.6) | 126.5 (7.8) | 105 (0) | 123 (20.7)
  systolic blood pressure after methamphetamine | 131.7 (15.5) | 114.3 (9.5) | 122 (4.2) | 131 (14.1) | 107 (0) | 119.7 (6.7)

ADVERSE EVENTS:
Time Frame: 8 hr
Arm/Group | Prazosin Effects on Methamphetamine
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin Effects on Methamphetamine (N=3)
hypotension (Vascular disorders) | 1 (1) — Orthostatic hypotension with prazosin 2 mg dose. BP 126/55 to 96/43 (sitting to standing); heart rate 118 to 95 (sitting to standing) dizziness, diaphoresis. Symptoms resolved with a 500 cc IV fluid bolus. No ectopy or ST segment changes were noted.

LIMITATIONS AND CAVEATS:
24 enrolled, 3 started study (1 withdrew after 5 sessions, 1 after 3 sessions; both for personal reasons), 1 completed. Data were collected on sessions completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes